CLINICAL TRIAL: NCT05765890
Title: Barriers to MASLD Management in Europe: Findings From a Multidisciplinary HCP-survey
Acronym: BARRIERS-MASLD
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: DAS-7671; U1111-1284-5875 (Other: World Health Organization (WHO))
Record Dates: First submitted 2023-02-14; First posted 2023-03-13 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Non-alcoholic Steatohepatitis (MASH); Non-alcoholic Fatty Liver Disease (MASLD)
MeSH Terms: conditions — Non-alcoholic Fatty Liver Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hepatologists: Recruited via email through online panel companies with which respondents have provided permission to be contacted for research purposes
  Interventions: Other: No treatment given
- Metabolically-Focused HCPs: Recruited via email through online panel companies with which respondents have provided permission to be contacted for research purposes
  Interventions: Other: No treatment given

INTERVENTIONS:
Other: No treatment given — No treatment given

SUMMARY:
The purpose of this study is to better understand the main barriers to earlier diagnosis and better management of MASLD/MASH patients and to understand the key barriers to adoption of guidelines.

This study is a cross-sectional design, conducted across 5 countries in Europe- France, Germany, Spain, United Kingdom (UK), Italy. Study participants, Hepatologists and other metabolically focused healthcare providers (HCPs), will be recruited to complete a 15 minute self-administered online survey.

ELIGIBILITY:
Inclusion Criteria:

For Hepatologists:

1. Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. Male or female, age above or equal to 18 years at the time of signing informed consent.
3. Is a physician
4. Lives in UK, France, Germany, Italy or Spain
5. Primary medical specialty is:

5.a. Hepatology or 5.b. Gastroenterology or Internal Medicine with a subspecialty in Hepatology 6. In practice at least 3 years 7. Spends at least 50 percent of their time in an office/clinic setting 8. Spends at least 60 percent of their time in direct patient care 9. Sees at least 15 patients/month with MASH/MASLD

For Metabolically-Focused HCPs (Endocrinologist/General Physician/Family Physician/Internal Medicine):

1. Informed consent obtained before any study-related activities (study-related activities are any procedure related to recording of data according to the protocol).
2. Male or female, age above or equal to 18 years at the time of signing informed consent.
3. Is a physician
4. Lives in UK, France, Germany, Italy or Spain
5. Primary medical specialty is:

5.a. General Physician/Family Practitioner or Endocrinology or 5.b. Internal Medicine without subspecialty in Hepatology 6. In practice at least 3 years 7. Spends less than 50 percent of their time in an office/clinic setting 8. Spends less than 60 percent of their time in direct patient care 9. Sees at least 15 patients/month with suspected/diagnosed MASH/MASLD 10. Sees and actively treats at least 30 patients/month with Type 2 Diabetes (T2D) and/or Obesity

Exclusion Criteria:

1. Previous participation in this study. Participation is defined as having given informed consent in this study
2. Mental incapacity, unwillingness or language barriers precluding adequate understanding or cooperation
3. Does not meet inclusion criteria requirements

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Hepatologists and other metabolically focused healthcare providers (HCPs)
Sampling Method: Non-Probability Sample
Enrollment: 675 (Actual)
Dates: Start 2023-03-24 (Actual); Primary Completion 2023-09-12 (Actual); Study Completion 2023-09-12 (Actual)

PRIMARY OUTCOMES:
Unaided awareness | At the time of survey response (Day 1)
  Open ended response
Aided awareness | At the time of survey response (Day 1)
  Multi- select from defined list
Behaviours relative to diagnosing and managing MASLD | At the time of survey response (Day 1)
  Numerical, multi-select from defined list
Use of current guidelines | At the time of survey response (Day 1)
  Multi-select from defined list; Likert scales; Numerical
  Likert scales:
  1=Not at all Relevant, 7=Extremely Relevant
Barriers in guideline adoption | At the time of survey response (Day 1)
  Multi-select from defined list; Likert scales; Numerical
  Likert scales:
  1=Doesn't impact at all, 7=Greatly impacts

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Transparency (dept. 2834), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Bangalore, India

IPD SHARING:
Plan to Share IPD: Yes
"According to the Novo Nordisk disclosure commitment on novonordisk-trials.com"
URL: http://novonordisk-trials.com